CLINICAL TRIAL: NCT00634894
Title: A Phase II, Double-Blinded, Randomized Evaluation of Femara (Letrozole) Versus Placebo for Adjuvant Treatment After Completion of First-Line Chemotherapy for Patients With Optimally Debulked and Chemoresponsive Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Femara (Letrozole) Versus Placebo for Patients With Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted with no registration, the drug company sponsor withdrew support.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-0689
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2009-09

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Femara; Letrozole; Placebo
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femara (Experimental)
  Interventions: Drug: Femara
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Femara — 2.5 mg by mouth daily x 12 weeks
  Other Names: Letrozole
  Arms: Femara
Drug: Placebo — Placebo capsule by mouth daily x 12 weeks
  Arms: Placebo

SUMMARY:
Primary Objective:

1. Evaluate the efficacy of letrozole to increase the duration of progression-free survival (defined as time to earliest occurrence of local or distant recurrence or clinically significant elevation in CA-125) when used as adjuvant treatment after completion of primary surgery and first line platinum containing chemotherapy in patients with optimally debulked (< 1 cm residual disease) stage IIA-IIIC ovarian, fallopian tube, or primary peritoneal cancer.

Secondary Objective:

1. Observe the incidence of local and distant recurrences.

DETAILED DESCRIPTION:
THE STUDY DRUG:

Letrozole is designed to block the enzyme that makes estrogen in post-menopausal women. By interfering with the production of estrogen made by the enzyme, letrozole decreases the total amount of estrogen in the body. As a result, less estrogen can reach cancer cells, which may prevent their growth.

SCREENING TESTS:

Before you can begin taking the study drug on this study, you will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed:

* Your complete medical history will be recorded.
* You will have a physical exam, including a pelvic exam and measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* Blood (about 2-3 teaspoons) will be drawn for routine tests and to test for tumor markers.
* You will have a chest x-ray and a computed tomography (CT) scan or magnetic resonance imaging (MRI) scan to check the status of the disease.
* Your previously collected tumor tissue, if available, will be tested to learn if the estrogen receptor is positive or negative.
* You will be asked how well you are able to perform the normal activities of daily living (performance status evaluation).

STUDY GROUPS:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Group 1 will take letrozole. Group 2 will take a placebo. A placebo is a substance that looks like the study drug but has no active ingredients. Neither the doctor nor you will know which group you will be in. However, if needed for your safety, the study staff and study doctor will be able to find out which group you are in.

STUDY DRUG ADMINISTRATION:

You will take letrozole or the placebo by mouth 1 time every day of each 12-week study "cycle". It should be taken around the same time every day and can be taken with or without food and/or water. You will be given the amount of study drug/placebo needed for 1 cycle of therapy at a time.

You will keep a drug "diary" during the study. In this diary you will list when and how much study drug/placebo you took. This diary will be reviewed after each cycle.

STUDY VISITS:

Within 4 weeks before your first dose of study drug/placebo, you will have a bone scan to test your bones and to watch for any signs of osteoporosis (weakened bones) that can be caused by decreased estrogen levels. You will be separately consented for this bone scan, which will describe the procedure and its risks in detail.

Every 12 weeks, the following tests and procedures will be performed:

* Blood (about 2-3 teaspoons) will be drawn for routine tests and to test for tumor markers.
* You will have a CT scan of the chest, abdomen, and pelvis to check the status of the disease.
* You will have a physical exam, including a pelvic exam and measurement of your vital signs and weight.
* You will have a performance status evaluation.
* You will be asked if you have experienced any side effects.

Every 6 months, you will have a chest x-ray.

Every year, you will have a bone scan to check for osteoporosis.

LENGTH OF STUDY:

You may remain on the study for as long as you are not experiencing intolerable side effects and the disease has not gotten worse. In that case, you will be taken off study. The total length of the study is five (5) years. At the end of the study, if you are still on active treatment, you and your doctor may or may not decide to continue treatment off-study.

END-OF-STUDY VISIT:

On the last day that you take the study drug/placebo, you will have an end-of-study visit. The following tests and procedures will be performed:

* Blood (about 2-3 teaspoons) will be drawn for routine tests and to test for tumor markers.
* You will have a physical exam, including a pelvic exam and measurement of your vital signs and weight.
* You will have an MRI scan or CT scan to check the status of the disease.
* You will have a performance status evaluation.
* You will be asked if you have experienced any side effects.

This is an investigational study. Letrozole is commercially available and FDA approved for the treatment of some types of breast cancer. Its use in patients with ovarian cancer is experimental. While you are on study, letrozole or the placebo will be provided at no cost to you.

Up to 50 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with optimally debulked (< 1 cm residual disease) stage IIA-IIIC ovarian, fallopian tube, or primary peritoneal cancer that have achieved a complete clinical response (CR) to first-line surgery and chemotherapy.
2. All patients must have had appropriate surgery with appropriate tissue available for histologic evaluation to confirm diagnosis and stage.
3. Patients must have completed primary treatment within the past 8 weeks and received at least 5 cycles and not more than 8 cycles of a platinum (IV or IP) and paclitaxel or docetaxel-based combination chemotherapy. Patients must have no symptoms suggestive of persistent cancer.
4. Patient must have a CT or MRI scan of the abdomen/pelvis with no evidence of metastatic disease and a normal CA-125 (< 35 Units/mL) following primary therapy.
5. Patients willing to sign informed consent to participate in study for 5 years or until first recurrence.

Exclusion Criteria:

1. Patients with any evidence of metastatic disease after completion of surgery and first line chemotherapy
2. Patients with low grade ovarian cancer histology.
3. If chemotherapy initiated greater than 8 weeks after primary surgery or completed more than 8 weeks prior to treatment start.
4. Patients that received neoadjuvant chemotherapy.
5. Patients taking any form of HRT and/or CAM products (i.e. phytoestrogens, etc.)
6. Patients with history of prothrombic clotting disorders (i.e PE or DVT).
7. Patients with history of malignant disease within past 10 years except for squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix, adequately cone biopsied
8. Patients with severe concomitant disease which would place patient at unusual risk or confound the results of the trial.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Median Progression-free survival (PFS): Time to progression or death from complete response (CR) | Assessed after 12 weeks of therapy, and followed for 36 months post-treatment
  PFS defined as time to earliest occurrence of local or distant recurrence or clinically significant elevation in CA-125. Biochemical progression is defined as two serially rising serum values of CA-125 greater than or equal to two times the upper limits of normal (ULN >35 U/ML) performed at least one week apart, regardless of CT scan results.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Wolf, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org